CLINICAL TRIAL: NCT00504634
Title: A Phase II Trial of Bortezomib (Velcade) After Allogenic Peripheral Blood Stem Cell or Bone Marrow Transplantation for Patients With Multiple Myeloma
Brief Title: Bortezomib (Velcade) Post Allogenic Peripheral Blood Stem Cell Transplantation for Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0751
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Post Allogeneic Transplantation; Bortezomib; Velcade; PS-341
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): 1 mg/m^2 intravenous (IV) Days 1, 4, 8, and 11.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 1 mg/m^2 IV On Days 1, 4, 8, and 11.
  Other Names: Velcade; PS-341

SUMMARY:
Primary Objective:

1. To determine the antimyeloma effect of bortezomib after allogeneic transplantation for patients with multiple myeloma.

Secondary Objective

1. To determine the toxicity profile of bortezomib in patients with multiple myeloma undergoing allogeneic progenitor cell transplantation.

DETAILED DESCRIPTION:
Bortezomib (velcade) is a new drug that works by blocking a structure in the cells called proteasome. This proteasome acts like a system that eliminates abnormal or old proteins from the cells. Cancer cells may be sensitive to drugs like bortezomib (velcade), because tumor cells have more abnormal proteins than normal cells. Bortezomib (velcade) enters the tumor cells and affects the way they divide. When cancer cells cannot divide, they die.

You will have blood (about 2 tablespoons) and bone marrow testing done about every 2-3 months to determine your response and tolerance to treatment. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle.

You will receive bortezomib (velcade) as an infusion into a vein over 5-10 minutes twice a week for 2 weeks. You will then rest for 10 to 17 days. This 21-28 day period makes up 1 cycle. You will complete up to a total of 4 cycles. Courses 2 and 3 might be given under supervision of your local physician however the principal investigator will do necessary treatment dose adjustments and new set of treatment orders will be provided to your physician. Treatment evaluations will be under the supervision of the principal investigator.

You will have a physical exam and routine blood tests (about 2 tablespoons) before each dose of bortezomib (velcade). Blood (about 2 tablespoons) and urine tests to determine response to treatment will be performed once a month, as well as blood tests to look at side effects of treatment, will be performed at least once a week and more frequently if medically necessary.

You will be taken off study if the disease gets worse or intolerable side effects occur. You will be called every 3 months for at least 1 year after the last dose of bortezomib (velcade) to see how you are doing.

This is an investigational study. Bortezomib (velcade) is commercially available and indicated for the treatment of myeloma. A total of 28 patients will participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma at least 3 months post allogeneic transplant who either failed to achieve a complete remission or are relapsing.
* Allograft performed from a related donor who is HLA-compatible (5/6 or 6/6), or class I serologic match and class II molecular matched unrelated donor).
* Zubrod Points Scale (PS) < 2, life expectancy is not severely limited by concomitant illness.
* Patient willing and able to sign informed consent.
* Patients less than 70 years of age.

Exclusion Criteria:

* Active Central Nervous System (CNS) disease.
* Uncontrolled acute or chronic Graft-versus-host disease (GVHD).

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Complete Response (CR) | 6 weeks from beginning treatment
  Response rate (CR), evaluated within 6 weeks of beginning treatment, assessed using The European Group for Blood and Bone Marrow Transplant/International Bone Marrow Transplant Registry (EBMT/IBMTR) response criteria of Complete Response (CR), Minimal Response (MR), No Change (NC), or Progressive Disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio A. Giralt, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org